CLINICAL TRIAL: NCT07006623
Title: A Multicenter Study of the Cognitive Model for Behavioral Interventions (CoMBI) as a Personalized Cognitive Behavioral Intervention for Patients With Severe Mental Illness
Brief Title: "CoMBI-SMI Multicenter Study: A Person-Centered Cognitive-Behavioral Intervention for Severe Mental Illness"
Acronym: CoMBI-SMI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Mondriaan (Unknown)
Responsible Party: Principal Investigator, Saskia Bollen, Hoofdonderzoeker, Vrije Universiteit Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METCZ20250033; projectnr 330 (Other Grant/Funding Number: Stichting tot Steun Nederland)
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Mental Illness Persistent
Keywords: Severe mental illness; older adults; adults; mediationtherapie; Cognitive behavioral therapie; Nursing interventions
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CoMBI-SMI (Experimental): This study arm includes adults (aged 18-64 years) and older adults (aged 65 years and older) with a severe mental illness (SMI). Participants must meet the inclusion criteria of having a diagnosed SMI and exhibiting behavior that is not well understood by caregivers. Additional inclusion criteria are the willingness and ability to participate in the study procedures. Participants in this arm will receive the CoMBI-SMI intervention following a period of treatment as usual.
  Interventions: Behavioral: CoMBI-SMI

INTERVENTIONS:
Behavioral: CoMBI-SMI — CoMBI-SMI (Cognitive Model for Behavioral Interventions - Severe Mental Illness) is a structured, team-based behavioral intervention for individuals with severe mental illness. It consists of four steps: (1) analyzing misunderstood behavior and identifying unmet core needs, (2) selecting the most relevant core need, (3) choosing appropriate nursing interventions, and (4) developing a CoMBI care plan. The model is based on cognitive-behavioral principles and personality-based formulations grounded in the DSM. It describes self-image, perception of others, triggers, and problematic behaviors. CoMBI-SMI is implemented by the entire team in a cyclical process, with periodic evaluation and a focus on consistent, team-aligned strategies.

SUMMARY:
This observational multicenter study aims to evaluate whether the Cognitive Model for Behavioral Interventions - Severe Mental Illness (CoMBI-SMI) can reduce challenging behaviors and psychological symptoms in adults (aged 18 and older) with severe mental illness (SMI). The study is conducted across multiple sites in the Netherlands, Belgium, and the Caribbean, using a stepped-wedge design. All participating departments initially continue their usual care. At different time points, each team receives training in the CoMBI-SMI approach and begins implementing the intervention. This design allows for a comparison between standard care and CoMBI-SMI-based care.

Participants first receive their usual treatment, during which baseline data are collected on their behavior and psychological symptoms. After the care team is trained in CoMBI-SMI, participants receive CoMBI-SMI-based care for four weeks. They complete questionnaires on behavior, psychological symptoms, and quality of life before and after the intervention. The study aims to assess whether CoMBI-SMI helps reduce challenging behaviors such as aggression or repetitive actions, improve quality of life, and reduce stress for both caregivers and treatment teams. Findings from this study may help improve care for individuals with severe mental illness and provide better support for mental health professionals managing complex behaviors.

DETAILED DESCRIPTION:
This multicenter observational study investigates the effectiveness of a treatment protocol for a personalized approach to behavioral problems in individuals with severe mental illness (SMI), grounded in patients' core psychological needs derived from their specific personality traits. Participants will be recruited from specialized mental health care institutions in the Netherlands, Belgium, and the Caribbean. Both adults (aged 18-64 years) and older adults (≥65 years) with SMI will be included.

The study employs a stepped-wedge design, where all participating teams initially provide treatment as usual (TAU), with outcome measurements every four weeks. At staggered time points, teams will be trained in the CoMBI-SMI intervention and transition to providing care based on this model. CoMBI-SMI (Cognitive Model for Behavioral Interventions - Severe Mental Illness) is a mediation-based approach in which behavioral interventions are implemented through a multidisciplinary team, rather than individual therapy. This model is particularly suited for the SMI population, where direct psychotherapy is often unfeasible due to lack of motivation or cognitive limitations.

The CoMBI-SMI intervention is based on Beck's cognitive model of personality disorders and integrates structured nursing interventions from the Nursing Interventions Classification (NIC). The intervention begins with the identification of maladaptive behavior patterns by the care team. These behaviors are analyzed in terms of their environmental triggers and maintaining consequences. A relevant core need is then selected from the CoMBI-SMI framework, and corresponding team-based interventions are planned. These are documented in a CoMBI care plan and implemented in a cyclical, evaluation-based format.

Primary outcome measures are the Neuropsychiatric Inventory Questionnaire (NPI-Q), assessing behavioral symptoms and associated distress, and the Brief Symptom Inventory (BSI), measuring psychological symptom severity. Secondary outcomes include perceived caregiver burden (NPI-Q distress scores) and patient-reported quality of life, measured by the Mental Health Quality of Life scale (MHQoL-7D). In addition, the study will identify predictive factors for treatment response using personality assessment tools: the Personality Inventory for DSM-5 - Brief Form + Modified (PID-5-BF+M) and the Level of Personality Functioning Scale - Brief Form 2.0 (LPFS-BF 2.0).

The NPI-Q data will also be used for a validation substudy in the SMI population, evaluating the instrument's construct validity, internal consistency, and inter-rater reliability.

Healthcare providers in participating departments will be trained in the CoMBI-SMI protocol. Training consists of an online theoretical module followed by a Meet-the-Expert (MTE) session, where providers can discuss theory and practice the application of CoMBI-SMI using clinical case studies. Completion of the training requires passing case-based assessments that evaluate theoretical understanding and clinical reasoning.

This study aims to improve behavioral management in SMI, enhance team competence in dealing with complex behaviors, and contribute to the development of structured, theory-based protocols for mediation therapy in psychiatry.

ELIGIBILITY:
Inclusion Criteria:

* Psychogeriatric inpatients aged 18 years and older
* Clinical diagnosis of a severe mental illness (SMI)
* Presence of behavioral problems not understood by caregivers
* Willingness and ability to participate in the study

Exclusion Criteria:

- Diagnosis of dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Neuropsychiatric Inventory - Questionnaire (NPI-Q): Symptom Severity and Caregiver Distress Scores | At baseline (before the start of treatment-as-usual) Immediately before the start of CoMBI-SMI training At week 5 (after 4 weeks of CoMBI-SMI-based care)
  The NPI-Q is a validated 12-item questionnaire used to assess neuropsychiatric symptoms and associated caregiver distress. The questionnaire is completed by an informal caregiver and evaluates whether specific symptoms are present, the severity of each symptom (rated on a 3-point scale from 1 = mild to 3 = severe), and the emotional distress it causes the caregiver (rated on a 6-point scale from 0 = not at all distressing to 5 = extremely distressing). Higher scores indicate more severe symptoms and greater caregiver distress. Total scores for symptom severity range from 0 to 36, and for caregiver distress from 0 to 60.
Brief Symptom Inventory (BSI): Total Symptom Severity Score | At baseline (before the start of treatment-as-usual) Immediately before the start of CoMBI-SMI training At week 5 (after 4 weeks of CoMBI-SMI-based care)
  The Brief Symptom Inventory (BSI) is a 53-item self-report questionnaire used to assess psychological and somatic symptom severity over the past week. Items are scored on a 5-point Likert scale ranging from 0 = "not at all" to 4 = "extremely." The instrument yields scores for nine subscales (Somatization, Cognitive Problems, Interpersonal Sensitivity, Depression, Anxiety, Hostility, Phobic Anxiety, Paranoid Ideation, and Psychoticism), as well as a Global Severity Index (GSI), which reflects overall symptom severity. Higher scores indicate more severe psychological distress. The GSI score ranges from 0 to 4.
  The BSI is validated for use in clinical and general populations and has been standardized for the Dutch language area, with norm data for men and women in both clinical and non-clinical samples.

SECONDARY OUTCOMES:
Mental Health Quality of Life (MHQoL-7D): Total Score and Visual Analogue Scale (VAS) | At baseline (before the start of treatment-as-usual) Immediately before the start of CoMBI-SMI training At week 5 (after 4 weeks of CoMBI-SMI-based care).
  The Mental Health Quality of Life (MHQoL-7D) is a standardized self-report instrument designed to assess quality of life in individuals with mental health conditions. It consists of two components: (1) the MHQoL-7D descriptive section, comprising seven dimensions (self-esteem, independence, mood, relationships, daily activities, physical health, and future), each scored on a 4-point scale from 0 = "very dissatisfied" to 3 = "very satisfied"; and (2) a visual analogue scale (VAS) that measures overall psychological well-being on a scale from 0 = "the worst imaginable psychological well-being" to 10 = "the best imaginable psychological well-being."
  Total scores on the MHQoL-7D range from 0 to 21, with higher scores indicating better quality of life. The VAS provides a single-item global rating of subjective mental health.

OTHER OUTCOMES:
Personality Inventory for DSM-5 - Brief Form Plus Modified (PID-5-BF+Modified): Domain Scores | Once, immediately before the start of CoMBI-SMI training
  The Personality Inventory for DSM-5 - Brief Form Plus Modified (PID-5-BF+Modified) is a 36-item self-report questionnaire derived from the original 220-item PID-5. It assesses maladaptive personality traits across six domains: Negative Affectivity, Detachment, Antagonism, Disinhibition, Psychoticism (from DSM-5), and Anankastia (from ICD-11). Items are scored on a 4-point Likert scale ranging from 0 = "very false or often false" to 3 = "very true or often true." Each domain score is calculated as the mean of its respective items.
  Higher scores indicate greater expression of maladaptive personality traits. Each domain score ranges from 0 to 3.
  The PID-5-BF+Modified will be used in both self-report and informant-report formats to explore associations between personality pathology and intervention outcomes.
Level of Personality Functioning Scale - Brief Form 2.0 (LPFS-BF 2.0): Total Score and Domain Scores | Once, immediately before the start of CoMBI-SMI training
  The Level of Personality Functioning Scale - Brief Form 2.0 (LPFS-BF 2.0) is a 12-item self-report questionnaire that assesses the severity of personality dysfunction, in line with Criterion A of the Alternative Model for Personality Disorders (DSM-5). It covers four domains of personality functioning: Identity, Self-Direction, Empathy, and Intimacy. Each domain is represented by three items. Items are scored on a 5-point Likert scale ranging from 0 = "completely false" to 4 = "completely true."
  Domain scores are calculated as the mean of the corresponding three items. The total score is the mean of all 12 items and ranges from 0 to 4. Higher scores indicate greater impairment in personality functioning.
  The LPFS-BF 2.0 will be administered in self-report and informant-report formats to assess baseline levels of personality dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: van Alphen, Prof. dr., Principal Investigator — Mondriaan
Locations (1):
- Mondriaan, Heerlen, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No